CLINICAL TRIAL: NCT01769859
Title: Systematic Genetic Analysis of Phenomenology and Treatment Response in Mood Disorders
Status: Terminated | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); The Cleveland Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Fan General; KL2TR000440 (NIH)
Record Dates: First submitted 2013-01-11; First posted 2013-01-17 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: Bipolar Disorder; Major Depressive Disorder; Genetics
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary goals of this work are: a) to establish a unique collection of mood disorder patients across the life cycle, including children, adults and geriatric patients, with well-defined medical co-morbidities and medication treatment outcomes at the University Hospitals Case Medical Center Department of Psychiatry; b) to establish a collection of nuclear families, including both mothers and fathers, of children diagnosed with mood disorders; c) to perform a systematic genetic analysis of the proposed sample repository to identify genes and genetic variants contributing to inter-patient variability in clinical phenotypes and treatment responses. Our primary hypothesis is that genetic variations may underlie individual variability in disease susceptibility, clinical phenotypes and treatment safety, tolerability, and effectiveness.

DETAILED DESCRIPTION:
The study entails a one-time blood draw that will be used to obtain phenotypic data and DNA of all eligible mood disorders patients, and their parents (if applicable), who are treated within the Psychiatry Department at University Hospitals Case Medical Center (UHCMC). In rare instances, if a participant is unable to cooperate with a blood draw, a saliva sample will be collected instead of drawing blood. All eligible participants will be diagnosed with bipolar disorder or major depressive disorder, or be a parent of a child diagnosed with bipolar disorder or major depressive disorder, and will be seen for the study visit at the Department of Psychiatry at University Hospitals of Cleveland, 10524 Euclid Avenue, Cleveland, OH, 44106. Required lab specimens will be collected at University Hospitals Laboratory Services or the Department of Psychiatry, and analyzed at UHCMC and Case Western Reserve University (CWRU) or at an NIH sponsored sequencing or genotyping laboratory.

DNA sample from eligible subjects will undergo whole genome genetic analysis using array-based genotyping or sequencing technologies. The clinical phenotypes, treatment response profiles and genotype data will be analyzed using single and multivariate analyses in order to identify genes and genomic regions contributing to inter-patient variability in disease susceptibility, clinical phenotypes and treatment responses. Alternatively, as sequencing costs decline continuously, the DNA samples may undergo targeted genomic region deep sequencing or whole genome sequencing analysis.

Any clinical patient, research participant or parent of a child patient, seven years and older, within the Department of Psychiatry will be targeted for enrollment. Eligible participants will be diagnosed with DSM-IV bipolar disorder (type I, II, or not otherwise specified) or DSM-IV major depressive disorder, as determined by an extensive clinical interview and the Mini-International Neuropsychiatric Interview-Plus (MINI-Plus) if applicable or will be a parent of a child diagnosed with bipolar disorder or major depressive disorder.

The primary phenotype definition for the genetic analyses proposed here is DSM-IV diagnosis (BD or MDD), phenotypic variables (comorbidities etc.), and treatment response, defined either continuously (change in symptom measures) or categorically (response/non-response), made on the basis of structured diagnostic instruments.

In summary, we expect the following types of phenotypic data (as shown in the attached minimum data set CRF) to be available for majority of participants:

* Demographic information including gender, age and ethnicity.
* Psychiatric diagnosis and history including age of onset and course of mood disorder etc.
* Family history of illness including psychiatric disorders, diabetes and cardiovascular diseases.

The additional clinical variables (from minimum dataset and clinical trials) may define mood disorder subtypes that are more genetically homogeneous and therefore more likely to reveal the influence of genes.

Once a participant has signed the informed consent form, a blood sample of approximately 4 teaspoons of blood, or a saliva sample of approximately half a teaspoon of saliva, will be collected for DNA extraction. The DNA samples will be linked with phenotypic data collected from the study participants. The blood draw or saliva collection and minimum data set questions are the only procedures that participants will need to complete once they decide to participate in the study. The informed consent form will specify that the demographic and diagnostic information used for this study will be taken from participation within another study or from the medical records of clinical patients; participants will not participate in this study if they do not provide consent to use their data retrospectively.

ELIGIBILITY:
Only clinical patients or research participants seen within the Department of Psychiatry at UHCMC will be approached for participation in this study.

Inclusion Criteria:

* Patients must give consent/assent to participate by signing and dating the Institutional Review Board approved written informed consent form prior to the initiation of any procedures for this study
* Patients must be diagnosed with Bipolar Disorder or Major Depressive Disorder or must be the parent of a child diagnosed with Bipolar Disorder or Major Depressive Disorder
* Patients must be at least 7 years old
* Patients must be willing to give a blood or a saliva sample
* Permission from guardian if participant in under 18

Exclusion Criteria:

* Patient is not diagnosed with Diagnostic and Statistical Manual-IV (DSM-IV) bipolar disorder, or Major Depressive Disorder
* Patient lacks the capacity to provide informed consent

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mood Disorders Program of University Hospitals Case Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identify genetic variations contributing to inter-patient variability in disease susceptibility | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Fan, PhD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland